CLINICAL TRIAL: NCT03591211
Title: Bio-psycho-social Pathways Underlying the Effects of Qigong Among Comorbid Depressed Elderly With Chronic Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: I-Shou University (Other); Fujian University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, TSANG Hector Wing-Hong, Professor and Head of Department of Rehabilitation Sciences, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 81173316-2
Record Dates: First submitted 2018-06-26; First posted 2018-07-19 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Chronic Disease; Depressive Symptoms
MeSH Terms: conditions — Chronic Disease; Depression | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qigong Training (Experimental)
  Interventions: Behavioral: Qigong Training
- Cognitive Training (Active Comparator)
  Interventions: Behavioral: Cognitive Training

INTERVENTIONS:
Behavioral: Qigong Training — Eight-Section Brocades; participants were trained individually.
  Arms: Qigong Training
Behavioral: Cognitive Training — Cognitive Training of Memory and Executive Function with Activities requiring Mobilization
  Arms: Cognitive Training

SUMMARY:
Depression and chronic medical conditions are common in older adults. Qigong is increasingly documented to have anti-depressive effects for older adults. Nevertheless, the scientific concepts behind qigong remain a mystery. To fill the knowledge gap, the neurobiological mechanism of the effects of qigong was explored. In addition, the benefits of qigong on subjective well-being, functional independence, sleep quality, mobility, and muscle strength were also tested. After random assignment, intervention group (n = 14) went through individual qigong exercise twice a week and for 12 weeks,whereas control group (n = 16) was involved in cognitive training activities with mobilization elements. The psychosocial, physical, and neurobiological outcomes of the two groups were compared.

ELIGIBILITY:
Inclusion Criteria:

* aged 60 or above
* have been suffering from chronic medical conditions for more than one year
* have depressive symptoms as indicated by Geriatric Depression Scale (GDS ≥ 6)

Exclusion Criteria:

* have practiced or received training of any form of mind-body exercises (including tai chi, yoga, and qigong) during the 6 months prior to intervention.
* have changed medication or the dosage prior to or during intervention
* have obvious cognitive and language impairment or score less than 20 in Mini-Mental State Examination (MMSE)
* undergo electroconvulsive therapy, psychotherapy, or psychoeducation
* cannot demonstrate satisfactory sitting balance

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ) | the change from baseline to the completion of intervention (12 weeks later)
  Patient Health Questionnaire (PHQ) is used to assess the experience of depressive symptoms. The frequency of each symptom was indicated based on a 4-point scale (0 = never; 3 = almost every day). A total score ranged from 0 to 27 can be derived, with higher score indicating severer depressive symptoms.

SECONDARY OUTCOMES:
Salivary Cortisol Level | baseline and 12 weeks after baseline
  measured with saliva sample obtained 5 times (07:00, 10:30, 13:00, 14:30, and 18:00) at two consecutive days at baseline and 12 weeks after baseline
Brain Deprived Neurotrophic Factor (BDNF) Level | baseline and 12 weeks after baseline
  measured with peripheral blood samples (10 ml) collected in the morning
Serotonin 5-HT Level | baseline and 12 weeks after baseline
  measured with serum extracted from blood samples. Around 2-3 ml of serum is harvested per 5 ml of blood.
Depression Anxiety Stress Scale (DASS-21) | baseline, 12 weeks after baseline, and 16 weeks after baseline
  Depression Anxiety Stress Scale (DASS-21) is a 21-item scale to measure symptoms of depression, anxiety, and stress with 7 items for each. Each item is measured with 4-point from 0 (never) to 3 (almost always). The scores of depression, anxiety, and stress are the sum of all subscale items, and it can range from 0 to 21. Higher score shows more severity of depression, anxiety, and stress.
Personal Well-Being Index (PWI) | baseline, 12 weeks after baseline, and 16 weeks after baseline
  It is measured by the 8-item scale of Personal Well-Being Index (PWI). Each item was rated according to an 11-point scale ranging from '0' (extremely dissatisfied) to '10' (extremely satisfied). An overall score of PWI score was the sum of all items. The overall score ranges from 0 to 110, with higher score indicating higher subjective well-being.
Functional Independence Measure (FIM) | baseline, 12 weeks after baseline, and 16 weeks after baseline
  It is measured by the 18-item scale of Functional Independence Measure (FIM). Based on a 7-point scale for rating (1
  = totally unable; 7 = totally independent), a total score of FIM ranges from 18 to 126 was generated. Higher total score indicates less disability.
Pittsburgh Sleep Quality Index (PSQI) | baseline, 12 weeks after baseline, and 16 weeks after baseline
  It is measured by the Pittsburgh Sleep Quality Index (PSQI). It has 19 items measuring 7 components of sleep quality, and a total score is calculated as the sum of all the component scores. The total score ranges from 0 to 21, with lower score showing better sleep quality.
Timed up and Go Test (TUG) | baseline, 12 weeks after baseline, and 16 weeks after baseline
  Timed up and Go Test (TUG) is used to measure mobility. During the test, participants were sitting on a chair, and then they were required to stand up, walk to a mark which is 3 meters away from the chair, go back to the chair from the mark, and sit down again. The time each participant spent to complete the above series of actions was recorded.
  Participants performed the test for three times, and their final scores were the average of the three. And lower score indicates better mobility.
Handgrip Strength | baseline, 12 weeks after baseline, and 16 weeks after baseline
  It is measured with a Jamar handheld dynamometer. Participants performed three trials of left hand and right hand grip strength, and the final outcome of each hand was calculated as the mean performance of the three trials. Higher score indicates stronger handgrip strength.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechinic University, Hong Kong, Hong Kong